CLINICAL TRIAL: NCT04113603
Title: Comparison of Diagnostic Performance of Urothelial Carcinomas Between Single-bolus and Split-bolus Computed Tomography Urography
Brief Title: Diagnostic Values of Urothelial Carcinomas: Single-bolus Versus Split-bolus Computed Tomography Urography
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Li-Jen Wang, Medical Imaging Department Director, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201701984A3
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A_Single bolus (Experimental): Single bolus computed tomography urography (CTU)
  Interventions: Diagnostic Test: Urinary malignancy
- B_Split bolus (Experimental): Split bolus computed tomography urography (CTU)
  Interventions: Diagnostic Test: Urinary malignancy

INTERVENTIONS:
Diagnostic Test: Urinary malignancy — Single bolus three phase CTU

SUMMARY:
Single-bolus computed tomography urography (CTU)is a recently developed one-stop imaging examination for diagnosis of urinary tract diseases, including urinary malignancies. However, single-bolus CTU uses two post- contrast phases (i.e.: nephrographic and excretory phases) for diagnosis of urinary tract diseases. A further-developed split-bolus CTU uses solitary post-contrast phase containing mixed information of nephrographic and excretory phases for diagnosis of urinary tract disease; however, whether split-bolus CTU has similar high diagnostic values for urinary malignancies remains unaddressed. Thus, the aim of this study is to compare the diagnostic performance between single-bolus and split-bolus CTU for diagnosing urinary malignancies. This study will enroll 352 patients from two hospitals if they fit the including criteria including aged > 40 years old, presenting with gross hematuria or having urinary malignancies histories, normal renal function (i.e.: estimated glomerular filtration rate > 60 mL/min/1.73 m2, no allergic history to iodinated contrast medium and no pregnancy). All enrolled patients will be randomized to undergo split-bolus and single-bolus CTU in 1: 1 manner. Two radiologists will read CTU images independently using a standardized recording sheet with Likert scales 1-5 representing higher probabilities of presence of urinary malignancies for larger number). The diagnostic values of split-bolus and single-bolus CTU will analyzed using reference standards by final diagnoses of urinary malignancies (i.e.: presence of urinary malignancies based on histological examinations of cytology examinations, biopsies or surgical specimens). The diagnostic performance of split-bolus CTU and single- bolus CTU for urinary malignancies will be compared using areas under receiver operating curve (ROC) to determine whether there is presence of significant difference .

DETAILED DESCRIPTION:
This study will enroll 352 patients. The calculation of sample size is according to the following equation:

n2=〖(Z∝+Zβ/2)〗^2/〖(δ-|ε|)〗^2 [p1(1-p1)/k+p1(1-p2)]

∝=0.05, β=0.2, δ=0.05, p1=0.96, p2=0.80 Then, the number of each arm patient should be ≥ 141 patients. However, if 20 % of the enrolled patients by fitting inclusion criteria are excluded by fitting exclusion criteria, the number of each arem should be ≥ 176 patients. Thus, this study plans to enroll 352 patients (for two arms). The enrolled patients are randomized to two groups (using single-bolus CTU versus using split-bolus CTU) using permuted block method.

ELIGIBILITY:
Inclusion Criteria: Fitting all of the followings

1. age ≥ 40 years old
2. presenting with gross hematuria or having a history of urothelial carcinomas
3. normal renal function (i.e.: estimated glomerular filtration rate ≧ 60 mL/min/1.73 m2)
4. no allergy history of iodinated contrast medium

Exclusion Criteria: Fitting any of the followings

1. pregnant or lactating woman
2. withdrawal of informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
diagnostic values of urothelial carcinoma | 3 years
  sensitivity, specificity, accuracy, area under ROC

SECONDARY OUTCOMES:
radiation dose | 3 years
  radiation dose of single bolus versus split bolus CTU

OTHER OUTCOMES:
diagnostic values of other urinary tract diseases | 3 years
  sensitivity, specificity and accuracy

CONTACTS AND LOCATIONS:
Overall Officials: Li-Jen Wang, M.D., M.P.H., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Li-Jen Wang, Taoyuan District, Ta, Taiwan

IPD SHARING:
Plan to Share IPD: No
Plan to make individual participant data